CLINICAL TRIAL: NCT07272902
Title: A Randomized Ablation-based Atrial Fibrillation Rhythm Control Versus Rate Control Trial in Patients With Heart Failure and Preserved Ejection Fraction (CABANA-RAFT HF): A Pilot Study
Brief Title: Treating Atrial Fibrillation in Heart Failure With Preserved Ejection Fraction: Ablation or Medication
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Ratika Parkash, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABANA-RAFT HF; 1032000 (Other: Nova Scotia Health REB File #)
Record Dates: First submitted 2025-11-24; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); Heart Failure With Mildly Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction (HFPEF); Rate Control; Rhythm Control
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Adrenergic beta-Antagonists; Calcium Channel Blockers; Digoxin

STUDY DESIGN:
Intervention Model Description: This trial is a pilot feasibility trial intended to lead into a larger, definitive trial as the trial is comparing two treatments already in clinical use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter Ablation (Rhythm Control Group) (Active Comparator): Participants in this group will undergo catheter ablation procedure, scheduled within 4 weeks of joining the study.
  Interventions: Procedure: Catheter Ablation for Atrial Fibrillation
- Medical Therapy (Rate Control Group) (Active Comparator): Participants in this group will take medications, with the dosages adjusted over the first few weeks to find the correct dosage.
  Interventions: Drug: Rate Control Medications (beta-blockers, calcium channel blockers, digoxin)

INTERVENTIONS:
Procedure: Catheter Ablation for Atrial Fibrillation — Participants randomized to this arm will undergo catheter ablation within 4 weeks of randomization. Pulmonary vein isolation is required; additional ablation strategies may be applied at investigator discretion. Guideline-directed medical therapy for atrial fibrillation and heart failure will also be provided.
  Arms: Catheter Ablation (Rhythm Control Group)
Drug: Rate Control Medications (beta-blockers, calcium channel blockers, digoxin) — Participants randomized to this arm will receive pharmacologic therapy to achieve guideline-recommended heart rate control (resting HR <80 bpm, <110 bpm with exercise). Therapy may include beta-blockers, non-dihydropyridine calcium channel blockers, or digoxin. If adequate control is not achieved with medication, AV nodal ablation and pacing may be used. Guideline-directed medical therapy for atrial fibrillation and heart failure will also be provided.
  Arms: Medical Therapy (Rate Control Group)

SUMMARY:
This study is testing two different ways of treating atrial fibrillation (AF) in people who also have heart failure with mildly reduced or preserved heart function. Patients will randomly be assigned to either rhythm control using catheter ablation or rate control using medicines. The pilot phase will determine if a larger study can be successfully carried out to see which approach better improves survival, reduces hospitalizations, and enhances quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of atrial fibrillation (documented on Holter, rhythm strip, or ECG)
* New York Heart Association (NYHA) class II-III heart failure
* Left ventricular ejection fraction (LVEF) >40%
* Meet specific NT-proBNP criteria:
* If HF hospitalization within 6 months prior to screening: NT-proBNP >200 pg/ml (if not in AF at screening) or >600 pg/ml (if in AF at screening)
* Otherwise: NT-proBNP >300 pg/ml (if not in AF at screening) or >900 pg/ml (if in AF at screening)
* On stable guideline-directed medical therapy for ≥1 month
* On stable diuretic dose for ≥2 weeks
* Suitable for either ablation-based rhythm control or rate control strategy

Exclusion Criteria:

* Permanent atrial fibrillation diagnosis
* Prior catheter ablation for atrial fibrillation
* NYHA class IV heart failure
* Rheumatic heart disease
* Moderate or severe mitral stenosis
* Mechanical mitral valve
* Severe aortic stenosis or severe aortic/mitral regurgitation
* Renal failure requiring dialysis
* Contraindication to oral anticoagulation
* Infiltrative cardiomyopathies
* Complex congenital heart disease
* Untreated thyroid disease
* Acute coronary syndrome or coronary artery bypass surgery within 12 weeks
* Participation in another clinical trial
* Inability to provide informed consent
* Other serious non-cardiovascular condition with life expectancy ≤1 year
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Trial Conduct | 12 months after randomization
  Recruitment rate (patients recruited per center per month) and crossover rate (percentage of participants switching study arms). Feasibility will be defined as ≥0.7 patients enrolled per center per month and ≤10% crossover.

SECONDARY OUTCOMES:
Composite of Cardiovascular Mortality and Heart Failure Hospitalization | Up to 12 months post-randomization
  Time to first event of cardiovascular death (due to MI, sudden cardiac death, HF, stroke, CV procedures, CV bleeding, or other CV cause) or hospitalization for heart failure (admission >24h, ED visit, or unscheduled IV diuretic administration).
All-Cause Mortality | Up to 12 months
  Death from any cause
Cardiovascular Hospitalizations and ED Visits (Non-HF) | Up to 12 months
  Number of hospitalizations or emergency department visits for other cardiovascular causes, including atrial fibrillation.
Quality of Life: EQ-5D (Euroquol 5D Questionnaire) | Baseline, 12 months
  EQ5D Will include responses from the Euroquol 5D questionnaire
Quality of Life: AFEQT (Atrial Fibrillation Effect on Quality of Life) Questionnaire | Baseline, 12 months
  AFEQT- Atrial Fibrillation Effect on Quality of Life Questionnaire (Scored 0-100, 0 is complete disability, 100 is no disability)
Quality of life- KCCQ-12 (Kansas City Cardiomyopathy Questionnaire-12) | Baseline, 12 months
  KCCQ-12- Kansas City Cardiomyopathy Questionnaire-12 (0-100, 0 is very poor, 100 is excellent)
Atrial Fibrillation Burden | Baseline, 3, 6, and 12 months
  Proportion of time in atrial fibrillation as measured by Holter monitoring and symptom-triggered ECG recordings
Change in NT-proBNP levels | Baseline, 12 months
  Change in plasma NT-proBNP levels from baseline to follow-up
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline, 12 months
  Change in LVEF as measured by echocardiography
Exercise Capacity (6-Minute Walk Distance) | Baseline, 12 months
  Change in distance walked in 6 minutes from baseline to follow-up
Recruitment Metrics | Throughout 12-month recruitment
  Recruitment ration of male vs. female participants, refusal rates and reasons.

OTHER OUTCOMES:
Procedural Complications | Up to 30 days post-ablation procedure
  Symptomatic pulmonary vein stenosis, atrio-esophageal fistula, pericardial effusion requiring pericardiocentesis, major bleeding requiring transfusion.
Antiarrhythmic Drug Adverse Events | Up to 12 months
  Incidence of drug-related toxicities (e.g., thyroid, hepatic, pulmonary, proarrhythmia)
All-Cause Death | Up to 12 months
  Number of deaths from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- QEII HSC, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No